CLINICAL TRIAL: NCT01628328
Title: Impact of Metallic Stent Insertion for Obstructing Colorectal Cancer on Circulating Tumor Cell Dissemination
Brief Title: Colonic Stent and Tumor Cell Dissemination
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: colonstent
Record Dates: First submitted 2012-06-21; First posted 2012-06-26 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Colorectal Cancer
Keywords: colonic stenting; colorectal cancer obstruction; circulating tumor cell
MeSH Terms: conditions — Colorectal Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stenting: patient who received colonic stenting for obstructive colorectal cancer
- Control: patients who had only colonoscopy without obstruction and without stenting

SUMMARY:
This study aims to examine the hypothesis of tumor cell dissemination after colonic stenting for obstructing colorectal cancer by measuring the level of plasma circulating tumor cell before and after the procedure of successful colonic stenting in patients.

DETAILED DESCRIPTION:
1. Patient recruitment:

   Patients will be recruited from the Division of Colorectal Surgery, Department of Surgery, the University of Hong Kong, over a 12 - 18 months period. Our institution is a tertiary referral center for colorectal cancer patients in Hong Kong. Informed consent will be obtained from the patients after the inclusion criteria are met.

   The study plans to recruit 25 patients in the colonic stenting group to compare with 15 patients in the control group.

   Inclusion criteria:

   Colonic stenting group
   1. Patients with obstructive colorectal cancer that requires colonic stenting as treatment
   2. Age > 18 years and is able to give informed consent
   3. Informed consent for blood collection obtained

   Control group
   1. Patients with colorectal cancer who have colonoscopy without stenting
   2. Age > 18 years and is able to give informed consent
   3. Informed consent for blood collection obtained
2. Blood collection and examination for circulating tumor cell

About 10ml of EDTA blood will be collected for examination before the procedure (colonoscopic stenting or colonoscopy in the control group) and blood collection daily will be repeated for 3 days after procedure. Blood will be sent to the laboratory for processing within 2 hours of withdrawal. Circulating tumour cells, which are characterized by CD45- (to exclude hematopoietic cells), CD326+ (to mark epithelial cells), CK18+ and CK19+ (to mark intestinal cells), i.e. cells expressing CD45-CD326+CK18/19+, will be detected by fluorescence activated cell sorting (FACS).

For each ml of blood, 1 ml of FCM Lysing solution will be added and allowed to incubate for 5 minutes to lyse the red blood cells, followed by centrifugation at 1000 RPM for 5 minutes. Supernatant will then be aspirated, and the pellet resuspend in approximately 1 ml cold 1X PBS. 10 µl of the appropriate antibody will be added into the tubes, vortexed and incubated for 15 in dark and room temperature. After incubation, cells will be washed with PBS and then incubated with the second antibody. The process is repeated until all 4 antibodies have been labelled to the cells. Cells will then be analysed on a FACS machine (MoFlo, Beckman Coulter).

ELIGIBILITY:
Inclusion Criteria:

* Colonic stenting group

  1. Patients with obstructive colorectal cancer that requires colonic stenting as treatment
  2. Age > 18 years and is able to give informed consent
  3. Informed consent for blood collection obtained

Control group

1. Patients with colorectal cancer who have colonoscopy without stenting
2. Age > 18 years and is able to give informed consent
3. Informed consent for blood collection obtained

Exclusion Criteria:

* Patients who refuse or who is unable to give informed consent on blood taking for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study plan to recruit 20-30 patients in the stenting group and about 10-20 patients in the control groups.
  There is no previous study on this topic and hence, no information availabe for statistical analysis of sample size required to show a difference.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Changes of circulating tumor cell level before and after colonic stenting for patients with obstructive colorectal cancer | Before and first 3 days after procedure
  The patients' peripheral blood will be collected before and on first 3 days after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jensen TC Poon, MS, Principal Investigator — Department of Surgery, University of Hong Kong